CLINICAL TRIAL: NCT06631365
Title: PrEPsmart Pilot: a Trial to Evaluate a Mobile App to Support the Safe and Effective Use of On-demand Pre-exposure Prophylaxis (PrEP) Among Sexual Minority Men in the US
Brief Title: PrEPsmart 2-1-1 Pilot
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-38355
Record Dates: First submitted 2024-08-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to the intervention (N=40) or control (N=20) conditions, using randomly-permuted blocks of randomly selected sizes 2 and 4, stratified by PrEP status (prescribed, non-prescribed). The randomization scheme will be generated and archived by the study statistician and implemented in RedCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- PrEPsmart intervention (N=40) (Experimental): Participants will be randomized in a 2:1 ratio to the intervention (N=40) For the pre-exposure prophylaxis (PrEP)smart intervention group, a study clinician will perform a medical history and limited physical exam to confirm eligibility to enroll in the study, a 4th generation rapid Human immunodeficiency virus (HIV) test will be performed, and labs drawn for creatinine, sexual transmitted infection (STI) testing (Neisseria gonorrhoeae/Chlamydia trachomatis (GC/CT)), syphilis), and hepatitis B testing.
  For participants newly starting 2-1-1 PrEP (PrEPsmart intervention group), study drug will be offered to participants to ensure that they will have access to PrEP during the study to be able to adequately test the app.
  Interventions: Device: PrEPsmart mobile app; Drug: Truvada
- control (N=20) (No Intervention): For the non-prescribed group, study staff will request documentation of an HIV-negative test within the last 3 months OR evidence of pre-exposure prophylaxis (PrEP) prescription within the last 6 months from medical records or pharmacy/provider communication. Additionally, study staff will confirm via self-report that the participant's 2-1-1 PrEP use will be clinically monitored by another clinician or clinic for the duration of the study. Any individual with a positive HIV test will have a confirmation test sent to the lab and be referred immediately for HIV care and initiation of treatment.
  For participants already on PrEP (control group) may choose to continue to use their own supply of Truvada (tenofovir disoproxil fumarate/emtricitabine, or TDF/FTC).

INTERVENTIONS:
Device: PrEPsmart mobile app — The PrEPsmart mobile app is an innovative and comprehensive app to support sexual minority men (SMM) using on-demand pre-exposure prophylaxis (PrEP) or daily PrEP. The PrEPsmart app consists of the following components:
  1. PrEP 211 dosing/sex diary and reminders
  2. Feedback on PrEP protection levels
  3. Quick tips
  4. Bi-directional secure messaging
  Arms: PrEPsmart intervention (N=40)
Drug: Truvada — Combination medication used in Human immunodeficiency virus (HIV) prevention, it blocks virus pathways to infection.
  Other Names: Emtricitabine; Tenofovir disoproxil fumarate
  Arms: PrEPsmart intervention (N=40)

SUMMARY:
This is a pilot study to assess the feasibility, acceptability, and preliminary effectiveness of pre-exposure prophylaxis (PrEP)smart among cisgender sexual minority males (SMM) taking on-demand PrEP over a 6-month period.

Upon project completion, the investigators will have developed a highly innovative tool to support men who have sex with men (MSM) using on-demand PrEP ready for testing in a larger efficacy trial

DETAILED DESCRIPTION:
This study is designed to enroll a diverse population of English-speaking cisgender sexual minority males (SMM) in the United States. The study team will enroll up to 60 participants who are taking or are interested in taking on-demand pre-exposure prophylaxis (PrEP). Participants will be randomized 2:1 to receive (intervention arm) or not receive (control arm) the PrEPsmart app at enrollment. Participants will complete follow-up visits at 3 and 6 months.

Participants newly starting 2-1-1 PrEP will be seen at the Bridge HIV clinic (prescribed group), while those already on PrEP may be seen at the clinic or complete visits virtually (non-prescribed group). Although no restrictions are put on the racial/ethnic make-up of the study participants, the site will strive to enroll at least 50% African American or Latino SMM into this study. The study will also strive to enroll at least 30% of participants who are newly starting or restarting 2-1-1 PrEP. Upon project completion, the study team will have developed a highly innovative tool to support men who have sex with men (MSM) using on-demand PrEP ready for testing in a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cisgender-male who reports sex with persons assigned male at birth
* Willing and able to provide written informed consent
* HIV-uninfected by negative 4th generation HIV test during screening (prescribed group)
* Documentation of negative HIV test within the last 3 months by outside laboratory OR evidence of PrEP prescription within the last 6 months based on medical records or pharmacy/provider communication
* Owns an iOS or Android mobile phone with a camera and has private access to the internet
* Able to understand, read, and speak English
* Able to attend study visits at a local research site in San Francisco (Bridge HIV) (prescribed and non-prescribed groups) or virtual visits via a HIPAA-compliant teleconferencing platform (non-prescribed group)
* Interested in starting or currently taking on-demand PrEP with TDF/FTC
* Report having anal sex at least once a month and expecting to maintain at least this frequency of anal sex during study participation by self-report
* Creatinine clearance ≥60 mL/min based on testing done during screening (prescribed group)
* Have PrEP clinical and laboratory monitoring by another provider or clinic by self-report (non-prescribed group)
* No contraindications to TDF/FTC use
* No evidence of chronic HBV infection based on testing done during screening (prescribed group)
* Willing to self-collect urine samples weekly

Exclusion Criteria:

* Repeatedly reactive HIV test at screening or enrollment or self-reported reactive HIV test (prescribed group)
* Signs or symptoms of acute HIV infection at screening or enrollment
* Currently enrolled in another PrEP intervention study.
* Unable to commit to study participation for the duration of the study
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender-male who reports sex with persons assigned male at birth
Enrollment: 60 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the PrEPsmart mobile app | 6 months
  Acceptability will be measured using the Client Satisfaction Questionnaire (CSQ-8) adapted for use in PrEPsmart pilot. The study team will also assess interest in future use of the app at study completion.
Usability of the PrEPsmart mobile app | 6 months
  Usability will be measured using the System Usability Scale (SUS) adapted for use in PrEPsmart pilot. A score >50 (out of 100) on the SUS indicates the app is acceptable.

SECONDARY OUTCOMES:
To compare PrEP coverage of sex acts as measured by weekly urine tenofovir test strips among SMM in the PrEPsmart vs. control arms | 6 months
  PrEP coverage will be primarily defined as self-reported sex acts in which the participant reported at least one pill taken within 24 hours before sex and one pill taken within 24 hours after sex, as defined in the Ipergay study. Additionally, the study team will conduct an analysis in which weekly PrEP dosing is confirmed by having a detectable TFV urine test within 7 days of reported sex.
To compare switching of PrEP regimens among SMM in the PrEPsmart vs. control arms | 6 months
  The proportion of participants who switch from on-demand PrEP to daily PrEP (or another regimen, e.g.
  injectable PrEP) will be calculated and compared between arms using chi-square tests.
To compare rates of PrEP discontinuation among SMM in the PrEPsmart vs. control arm | 6 months
  PrEP discontinuation and retention rates will be calculated, with 95% binomial confidence intervals, and compared between arms using log-binomial models. The study team will also estimate and compare time to discontinuation using Kaplan Meier methods and the log-rank test, accounting for censoring by end of study or dropout.
Elicit feedback on areas for improvement for PrEPsmart to guide further app refinement | 6 months
  Ideas for improvement of PrEPsmart elicited through exit interviews will be tabulated, discussed with the protocol team, and prioritized for development.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, Principal Investigator — albert.liu@sfdph.org
Locations (1):
- Bridge HIV, San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes